CLINICAL TRIAL: NCT06691828
Title: A Phase 1, Open-Label, 2-Period, Fixed-Sequence Study to Assess the Absolute Bioavailability, Absorption, Metabolism, Excretion, and Mass Balance of [14C]-NX-5948 in Healthy Males
Brief Title: Absolute Bioavailability, Absorption, Metabolism, Excretion, and Mass Balance Study of [14C] NX-5948
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nurix Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NX-5948-303
Record Dates: First submitted 2024-11-01; First posted 2024-11-15 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Active Treatment Arm IV and Oral (Experimental): This single Arm will include a single dose by IV and a single dose given by mouth for all 8 subjects.
  Interventions: Drug: NX-5948

INTERVENTIONS:
Drug: NX-5948 — NX-5948 will be given once by IV and then given once by mouth.

SUMMARY:
This is a Phase 1, 2-period, open-label, single-dose, fixed-sequence study to assess the absolute bioavailability, absorption, metabolism, excretion, and mass balance of [14C]-NX-5948. Period 1 will analyze PD (pharmacodynamics) and exploratory biomarkers. Period 2 will analyze total radioactivity and metabolite profiling.

DETAILED DESCRIPTION:
In Period 1 all subjects will receive a single dose of NX-5948 by IV and undergo pre and post dose labs to assess PK (pharmacokinetics) and PD parameters.

In Period 2 all subjects will receive a single dose of NX-5948 by mouth. Pre and post dose blood, urine, and feces will be collected until NX-5948 is no longer identified in samples.

Periods 1 and 2: Safety will be monitored throughout the study by repeated clinical and laboratory evaluations.

ELIGIBILITY:
Key Inclusion Criteria:

Subjects must fulfill all of the following inclusion criteria to be eligible for participation in the study:

* Healthy, adult, male, 18-55 years of age
* Subjects must follow protocol-specified contraception guidance as described in the protocol.
* Continuous non-smoker who has not used nicotine-and tobacco-containing products for at least 3 months prior to the first dosing based on subject self-reporting.
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2 at the screening visit.
* Medically healthy with no clinically significant medical history, physical examination, clinical laboratory profiles, vital signs, and 12-lead safety ECGs, at the screening visit and/or first check-in, as deemed by the PI or designee,
* Understands the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol.

Key Exclusion Criteria:

Subjects must not be enrolled in the study if they meet any of the following criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
* Clinically significant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neoplastic (including leukemia, lymphoma, malignant melanoma), myeloproliferative, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine or connective tissue diseases or disorders, or any illness that, in the opinion of the PI or designee, might confound the results of the study or pose an additional risk to the subjects by their participation in the study.
* History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing.
* History or presence of hypersensitivity, angioedema, or idiosyncratic reaction to the study drug(s) or related compounds.
* History or presence of:

  * Significant multiple and/or severe allergies, including anaphylactic reaction.
  * Personal or family history of prolonged QT syndrome or family history of sudden cardiac death.
  * Evidence of atrial fibrillation, atrial flutter, complete bundle branch block, Wolff-Parkinson-White Syndrome, or cardiac pacemaker.
  * Adrenal insufficiency.
  * Skin infection.
  * Any significant (as determined by the PI) drug-related allergic reactions such as, anaphylaxis, Stevens-Johnson syndrome, urticaria or multiple drug allergies.
* Has tattoo(s) or scarring at or near the site of IV injection or any other condition which may interfere with IV injection site examination, in the opinion of the PI or designee.
* Previous exposure to NX-5948.
* Any significant acute illness within 30 days prior to first dosing.
* Regular alcohol consumption > 14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine) prior to first dosing.
* Positive urine drug or alcohol results at the screening visit or first check in.
* Positive Coronavirus disease 2019 (COVID-19) results at first check-in.
* Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) at the screening visit.
* Has received radiolabeled substances or has been exposed to radiation sources over the past 12 months or is likely to receive radiation exposure or radioisotopes within the next 12 months such that participation in this study would increase their total exposure beyond the recommended levels considered safe (i.e., weighted annual limit recommended by the FDA 21CFR361 of 5000 mrem).
* Participation in another clinical study within 30 days or within 5 half-lives (if known), prior to the first dosing, whichever is longer. The 30-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study will enroll male subjects only.
Enrollment: 8 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Characterize Area Under the Curve (AUC0-inf), Half-life (T1/2) after IV dosing of NX-5948 | 9 weeks
  Characterize the Area Under the Curve (AUC0-inf), Half-life (T1/2) of a single IV dose of NX-5948 in healthy adult male subjects.
Evaluation of metabolite after oral dosing with [14C]-NX-5948 | 9 weeks
  Identify major metabolite and its AUC in plasma following a single oral dose of [14C]-NX-5948 in healthy adult male subjects.
Assessment of bioavailability with oral dosing of NX-5948 | 9 weeks
  Determine the absolute bioavailability (ABA) of an oral formulation of [NX-5948C]- in healthy adult male subjects.
Assessment of total radioactivity after oral dosing with NX-5948 | 9 weeks
  Determine the recovery of total radioactivity (TRA; mass balance) as a percentage of the administered dose after a single oral dose of [14C]-NX-5948 in healthy adult male subjects.
Assessment of whole blood to plasma ratio for TRA after oral dosing with NX-5948 | 9 weeks
  Characterize whole blood to plasma ratio for TRA following a single oral dose of [14C]-NX-5948 in healthy adult male subjects (i.e., whole blood:plasma partitioning ratio).
Characterize the Clearance (CL) after IV dosing of NX-5948 | 9 weeks
  Character the Clearance (CL) after IV dosing of NX-5948in healthy adults male subjects.
Characterize the Volume of distribution (Vz) after IV dosing of NX-5948 | 9 weeks
  Character the Volume of distribution (Vz) after IV dosing of NX-5948in healthy adults male subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Injac, MD PhD, Study Director — Nurix Therapeutics, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No